CLINICAL TRIAL: NCT07067710
Title: Effectiveness of Combined Motor Imagery and Action Observation in Improving Pain, Range of Motion, and Upper Limb Lymphedema in Breast Cancer Survivors. Efectividad de Las Terapias de imaginería Motora y observación de la acción en la Mejora Del Dolor, la Movilidad y el Linfedema de la Extremidad Superior en Supervivientes de cáncer de Mama.
Brief Title: The Use of Combined Motor Imagery and Action Observation to Evaluate the Influence on Functional Parameters Such as Strength, Range of Motion, Pain or Fear of Movement Among Others, in Females Breast Cancer Survivors.
Acronym: IM-OA23
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Miguel Servet (Other)
Collaborators: Instituto de Investigación Sanitaria de Navarra (IdiSNA) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PI_2023/81 Programa IM-OA23; PI_2023/81 (Other Grant/Funding Number: Department of Health of the Government of Navarra, Spain.)
Record Dates: First submitted 2025-01-09; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer Survivor
Keywords: Motor imagery; Action observation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMOA group (Experimental): The intervention group will participate in the IM-OA23 programme; the combination of motor imagery and action observation therapies.
  Interventions: Other: Motor imagery combined with action observation
- Control group (No Intervention): The control group will follow the usual care from primary care. There are no care programmes for long term cancer survivors.

INTERVENTIONS:
Other: Motor imagery combined with action observation — To observe and imaging one action with a video resource. Not virtual reality.
  Arms: IMOA group

SUMMARY:
The aim of this study is to evaluate the effectivity of the combined motor imagery and action observation therapies to improve functional parameters such as strenght, range of motion, pain or fear of movements among others in relation to upper limb in breast cancer survivors. The main question it aims to answer is: Will a combined therapy of motor imagery and action observation improve the strenght, rang of motion, pain, limb diameter and fear of movement of the upper limb in breast cancer survivor females? The participants will be part of the IM-OA23 proyect that consist on seeing some diferent videos about upper limb mobility and then they'll have to imagine the movements and to performed themselves. Researches will compare two groups (control group and intervention group) to evaluate the diferences between them.

DETAILED DESCRIPTION:
Purpose: The aim of this study is to evaluate the effectivity of a combined motor imagery and action observation protocol at strength, range of motion, limb diamter, and fear of movement of the upper limb of breast cancer survivors.

Methods: A randomised controlled clinical trial will be conducted. Subjects will be randomly assigned to the two randomly assigned to the two treatment groups: intervention (IM-OA23 programme) and control group (usual care).

This study will have pre and post measurements. The intervention consist on a display of diferent videos of upper limb movements and at daily living activities and in a excercise of imagine and doing this movements. The're will be used diferent tools such as a dynamometer, a goniometer, Visual Analogue Scale (VAS) of pain, or TSK questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Female, over 18 years, have suffered breast cancer, have ended active treatments (chemotherapy, radiotherapy, surgery), have pain or functional limitation or lymphedema at upper limb afected.

Exclusion Criteria:

* males, people with active treatments ongoning, other types of cancer, recurrence or metastasis of cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Sthrength | From enrollement to the end of the treatment at 6 weeks and 3 month after
  The grip strength of the hand of the affected limb shall be studied, using a dynamometer.
Range of Motion | From enrollement to the end of the treatment at 6 weeks and 3 month after
  The measurement of the degrees of movement of the shoulder joint by means of a goniometer. The movements of flexion, abduction and internal and external rotation shall be studied using previously established reference points.
  external rotation, using previously established reference points
Pain intensity | From enrollement to the end of the treatment at 6 weeks and 3 month after
  Pain intensity will be measured by Visual Analogue Scale (VAS). Participants will have to score their pain on a range from 0 to 10 where 0 means "no pain at all" and 10 "my pain is as bas as it could possibly be".
Limb diameter | From enrollement to the end of the treatment at 6 weeks and 3 month after
  Limb diameter will be measured by a measuring tape. The measurement is taken at the midpoint between the acromion and the olecranon, the tape being perpendicular to the limb without compressing the area. The midpoint is located with an elbow flexion of 90 degrees and then the measurement is taken with the elbow in extension, the result is expressed in centimetres.
Fear of movement | From enrollement to the end of the treatment at 6 weeks and 3 month after
  Fear of movement will be measured by the TSK questionnaire
Imagery | From enrollement to the end of the treatment at 6 weeks and 3 month after
  Imagery will be assessed using the Movement Imagery Questionnaire revised second edition (MIQ-RS)

CONTACTS AND LOCATIONS:
Overall Officials: Paula Escalada-Hernández, PhD, Study Director — Public University of Navarra; Nelia Soto-Ruiz, PhD, Study Director — Universidad Pública de Navarra; Pilar Arnal-Vallés, Candidate PhD, Principal Investigator — Hospital of Navarra
Locations (1):
- Public University of Navarre, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: Undecided